CLINICAL TRIAL: NCT01762345
Title: A Pilot Clinical Study of the Efficacy and Safety of a Disposable Intravaginal Device for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012099
Record Dates: First submitted 2012-12-12; First posted 2013-01-07 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary incontinence; SUI
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Pessaries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pessary device (Experimental): pessary (disposable intra-vaginal device)
  Interventions: Device: pessary (disposable intra-vaginal device)

INTERVENTIONS:
Device: pessary (disposable intra-vaginal device) — pessary device(disposable intra-vaginal device)manufactured by Procter & Gamble

SUMMARY:
This pilot study will evaluate the efficacy of the pessary (disposable intra-vaginal device) by reduction in urine leakage in women with stress urinary incontinence (SUI).

ELIGIBILITY:
Inclusion Criteria:

* have a ≥ 3 month history of experiencing Stress Urinary Incontinence
* be willing to use the pessary investigational device to control stress incontinence

Exclusion Criteria:

* pregnant, lactating or planning to become pregnant during the study
* within 3 months post partum
* intrauterine device (IUD) placement of less than 6 months
* a history of Toxic Shock Syndrome (TSS) or symptoms consistent with TSS
* experience difficulty inserting or wearing an intra-vaginal device, including a tampon
* vaginal surgery, perineal surgery, uterine surgery, or abortion (spontaneous or induced) within the past 3 months
* has any Screening laboratory value outside the laboratory reference range considered clinically significant by the Investigator
* for any reason, the Investigator decides that the subject should not participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Severance, MD, Principal Investigator — Radiant Research, Inc.
Locations (1):
- Study Center, Chandler, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 148 subjects entered the 2-week baseline phase and 65 dropped/failed before treatment
Period: Overall Study
Arm/Group | Pessary Device
Started | 83
Completed | 76
Not Completed | 7
Not completed — Adverse Event | 5
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pessary Device
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Pad Weight Gain
Description: Change from baseline as measured as reduction (improvement) in pad weight gain. Positive values are indicative of efficacious outcome.
Time Frame: from the 14-day baseline period to the last 7 days of 14-day device usage period
Population: Intent-to-Treat (ITT) population. The "Number of Participants Analyzed" is the number subjects with available (non-missing) data in week 2
Measure: Median (Inter-Quartile Range); unit: grams/usage period
Arm/Group | Pessary Device
Number analyzed (Participants) | 76
grams/usage period | 2.67 [0.12 to 12.7]

2. Primary Outcome: Change in Stress Urinary Incontinence Episodes
Description: Change from baseline as measured as reduction (improvement) in stress urinary incontinence episodes. Positive values are indicative of efficacious outcome.
Time Frame: from the 14-day baseline period to the last 7 days of 14-day device usage period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: episodes/usage period
Arm/Group | Pessary Device
Number analyzed (Participants) | 76
episodes/usage period | 0.92 [0.22 to 1.93]

3. Secondary Outcome: Change in Pad Weight Gain
Description: as for outcome 1
Time Frame: from the 14-day baseline period to the first 7 days of 14-day device usage period
Population: Intent-to-Treat (ITT) population. The "Number of Participants Analyzed" is the number subjects with available (non-missing) data in week 1
Measure: Median (Inter-Quartile Range); unit: grams/usage period
Arm/Group | Pessary Device
Number analyzed (Participants) | 82
grams/usage period | 2.36 [0.16 to 11.7]

4. Secondary Outcome: Change in Stress Urinary Incontinence Episodes
Description: as for outcome 2
Time Frame: from the 14-day baseline period to the first 7 days of 14-day device usage period
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: episodes/usage period
Arm/Group | Pessary Device
Number analyzed (Participants) | 82
episodes/usage period | 0.65 [0.17 to 1.66]

5. Secondary Outcome: Change in Quality of Life as Measured by Incontinence Impact Questionnaire (IIQ-7)
Description: The IIQ-7 is based on 7 questions referring to areas which may have been influenced or changed by accidental urine loss and/or prolapse. These questions are assigned a value of, 0 = 'Not at all,' 1= 'Slightly,' 2 = 'Moderately,' or 3 'Greatly.' The IIQ-7 is scored by taking the average score of items and then multiplying the average by 33 1/3 to put scores on a scale from 0 to 100. A lower score is considered less impact to quality of life and a higher score reflects more impact to quality of life. In the same manner, a reduction in scores from baseline reflects improved quality of life.
Time Frame: baseline and end-of-treatment
Population: Intent-to-Treat (ITT) population. The "Number of Participants Analyzed" is the number subjects with available (non-missing) data at the end of treatment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pessary Device
Number analyzed (Participants) | 82
units on a scale | 9.52 [0 to 28.6]

6. Other Pre Specified Outcome: Percentage of Responders for Pad Weight Gain
Time Frame: from the 14-day baseline period to the last 7 days of 14-day device usage period
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Pessary Device
Number analyzed (Participants) | 83
percentage of subjects | 36.6

7. Other Pre Specified Outcome: Percentage of Responders for SUI Episodes
Time Frame: from the 14-day baseline period to the last 7 days of 14-day device usage period
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Pessary Device
Number analyzed (Participants) | 83
percentage of subjects | 42.7

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: All adverse events reported by the subject from study initiation [Visit 1 (Screening)] until study completion [Visit 3 (End-of-Treatment)] were recorded.
Arm/Group | Pessary Device
Serious Adverse Events (participants affected / at risk) | 0/83
Other Adverse Events (participants affected / at risk) | 15/83
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pessary Device (N=83)
urinary tract infection (UTI) (Infections and infestations) | 5 (5) — UTI
vaginal hemorrhage (Reproductive system and breast disorders) | 5 (5) — vaginal bleeding
vaginal discomfort (Reproductive system and breast disorders) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The STUDY SITE and PRINCIPAL INVESTIGATOR agree that all data, calculations, interpretations, opinions and recommendations regarding the STUDY (hereinafter referred to as "RESULTS") shall be the property of P&G. The STUDY SITE and PRINCIPAL INVESTIGATOR agree to consider the RESULTS as INFORMATION subject to confidentiality restrictions